CLINICAL TRIAL: NCT02378987
Title: The Follow Study of Speech Functions in Preschool Children With Cerebral Palsy: Clinical Measures and Acoustic Analysis
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 99-1917B
Record Dates: First submitted 2015-02-25; First posted 2015-03-04 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2010-08

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; language; acoustic; motor speech; follow-up
MeSH Terms: conditions — Cerebral Palsy; Language

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Typical developmental children: Normal children
- CP children with GMFCS level I and II: Children with CP were classified into Levels I-II based on the Gross Motor Function Classification System (GMFCS).
- CP children with GMFCS level III and IV: Children with CP were classified into Levels III-IV based on the Gross Motor Function Classification System (GMFCS).

SUMMARY:
The aims of this study:

1. to investigate the difference in motor speech functions among children with cerebral palsy (CP) of different motor severities.
2. to investigate the longitudinal in motor speech functions at 6 months follow-up phase among children with CP of different motor severities.
3. the correlation between motor severity, personal factors, family factors, language ability and motor speech in children with CP.
4. to identify the variables that can predict motor speech functions in children with CP.

DETAILED DESCRIPTION:
Mental impairment, language and speech disorders are the common associated problems in children with CP. Previous studies focus on language and motor speech dysfunctions in children with CP at school-age child, adolescents and adults. Few literatures identify the determinants for predicted the motor speech performance in these children. It is important issue to follow-up the language and motor speech functions in children with CP. These data will provide clinicians for outcome prediction and goal setting.The aims of this study: (1) to investigate the difference in motor speech functions among children with CP of different motor severities, and(2) to investigate the longitudinal in motor speech functions at 6 months follow-up phase among children with CP of different motor severities, and(3) the correlation between motor severity, personal factors, family factors, language ability and motor speech in children with CP, and(4) to identify the variables that can predict motor speech functions in children with CP.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between the ages of 4-8 years old children.
2. Subjects which aged 7 years or older should sign a consent form by themself.
3. In line with the assessment, the case must be able to follow simple verbal commands, and can be done in a simple sentence description.
4. were diagnosed with spastic cerebral palsy.

Exclusion Criteria:

1. physiological condition is unstable: Included in three months for surgery or infection and other major diseases
2. there is progressive or degenerative symptoms or diseases (such as degenerative epilepsy), peripheral nerve injury, spinal cord injury.
3. visual perception or hearing problems, after correction difficult communicators.
4. other movement disorders patterns for children with cerebral palsy (athetoid type, offset type, etc.).

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children with CP having language ability greater than 3 years
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change of Peabody Picture Vocabulary Test-Revised | baseline and six months
  Children with CP underwent the assessments of Peabody Picture Vocabulary Test-Revised.

SECONDARY OUTCOMES:
Change of Percentage of Correct Consonant in six months | baseline and six months
  Children with CP underwent the assessments of Percentage of Correct Consonant

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, PhD, Principal Investigator — Department of Physical Medicine & Rehabilitation, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan